CLINICAL TRIAL: NCT06852872
Title: The Effect of Diathermy Therapy on Isolated Lumbar Extension (ILEX) Training
Acronym: ILEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences and Arts of Southern Switzerland (Other)
Responsible Party: Principal Investigator, Ron Clijsen, PhD., University of Applied Sciences and Arts of Southern Switzerland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-02308_ILEX
Record Dates: First submitted 2024-05-07; First posted 2025-02-28 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Resistance Training; Healthy Participants Study
Keywords: Isolated lumbar extension training; lumbar muscle; Thermal Therapy

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Investigator
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Capacitive Resistive Electric Transfer (CRET) therapy AND Isolate Lumbar Extension (ILEX) Training.
  Interventions: Other: CRET Therapy; Other: ILEX training
- Sham Group (Sham Comparator): Sham Capacitive Resistive Electric Transfer (CRET) therapy AND Isolate Lumbar Extension (ILEX) Training.
  Interventions: Other: ILEX training; Other: CRET therapy sham

INTERVENTIONS:
Other: CRET Therapy — Diathermy therapy with a protocol to preheat the back extensor muscle
  Other Names: TECAR therapy; Diathermy therapy
  Arms: Intervention group
Other: ILEX training — Isolated lumbar Extension Training
Other: CRET therapy sham — Diathermy therapy withouth any radiofrequency as a sham intervention
  Other Names: TECAR therapy; Diathermy therapy
  Arms: Sham Group

SUMMARY:
To evaluate the effectiveness of the Isolated Back Extension (ILEX) machine Myosom and examine the influence of preheating on resistance training, the investigators will recruit a cohort of 14 healthy individuals, including both male and female participants, who have no prior experience with ILEX training, for a 9-week training program consisting of a total of 18 sessions. Baseline (BL) measurements will be conducted in the week before the initiation of training, and two follow-up measurements (F/U 1 and F/U 2) carried out after the ninth and eighteenth sessions, with a minimum break of 48 hours after the last training session to ensure proper recovery and to prevent inaccuracies in muscle thickness measurement arising due to acute oedema.

DETAILED DESCRIPTION:
To evaluate the effectiveness of the Isolated Back Extension (ILEX) machine Myosom and examine the influence of preheating on resistance training, the investigators will recruit a cohort of 14 healthy individuals, including both male and female participants, who have no prior experience with ILEX training, for a 9-week training program consisting of a total of 18 sessions. Baseline (BL) measurements will be conducted in the week before the initiation of training, and two follow-up measurements (F/U 1 and F/U 2) carried out after the ninth and eighteenth sessions, with a minimum break of 48 hours after the last training session to ensure proper recovery and to prevent inaccuracies in muscle thickness measurement arising due to acute edema.

At BL, participants will need to give written informed consent and be familiarized to the back extensor machine and Category-Ratio-Scale (CR10) for the assessment of perceived effort and discomfort as well as thermal sensation and thermal comfort. Baseline assessment will include epidemiological data such as age, sex, height, and weight. At all three measurements (BL, F/U 1, F/U 2), the lumbar extensor musculature thickness (M. erector spinae) is evaluated through the ultrasound system Mylab2 (Esaote, Maastricht, Netherlands), the lower back flexibility is examined using a sit-and-reach test, and the isometric back extension endurance is measured through the Biering-Sørrensen test. Finally, maximal range of motion (ROM) and maximal voluntary isometric contraction will be evaluated using the Myosom machine.

Participants will be randomly assigned to either the sham group, which will receive a 10-minute treatment with Tecar device (T-Plus, Wintecare SA, Chiasso, Switzerland) turned off and not sending radiofrequency before each exercise session, or the intervention group, which will undergo a 10-minute treatment with the Tecar device to induce 448kHz capacitive monopolar radiofrequency and facilitate warming up of deep tissues. After every treatment the participants will be asked to rate their thermal sensation and comfort. Skin temperature will be measured using an infrared thermal imaging (FLIR A615 series, Emitec Industrial, Rotkreuz, Switzerland) after the first and final Tecar treatment.

Training will take place twice a week, beginning with a dynamic warm-up of the lumbar extensor for 120s, followed by three sets of resistance training (RT) lasting 120s, 120s, and 150s respectively, and concluding with a final set of dynamic recovery lasting 60s. 30-second recovery will be provided between every set. A low load will be used for the warm-up and recovery. The load will be subsequently increased until volitional fatigue. Repetitions will be executed by taking three seconds from complete flexion to complete extension, ensuring standardization at 20 repetitions per minute. A metronome with 40 beats per minute will provide audible feedback. The Myosom machine emits an audible signal upon completion of each phase of the repetition to guarantee a complete range of motion is achieved. Subsequent to every training session, participants will be requested to provide their effort (RPE-E) and discomfort (RPE-D) values.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* pain-free
* sufficient understanding of the German language
* able to give informed consent
* between 18 and 30

Exclusion Criteria:

* pregnant
* medication
* surgery of lumbar spine
* knee or hip disorders
* low back pain
* pathologies or deformities of lumbar spine
* other disorders
* previous or current ILEX Training

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
maximal isometric force of the back extensors | base line, 3 weeks, 6 weeks
  measured on the ILEX machine in Newton

SECONDARY OUTCOMES:
isometric back extension endurance | base line, 3 weeks, 6 weeks
  Biering- Sørensen test
Thickness of the Mm. erector spine | base line, 3 weeks, 6 weeks
  Ultrasound
Lumbar flexibility | base line, 3 weeks, 6 weeks
  Sit and reach test
Lumbar R.O.M. | base line, 3 weeks, 6 weeks
  ILEX machine
rating of perceived effort | After each of the 12 training sessions, twice a week for 6 weeks
  Category Ratio Scale (0-10)
rating of perceived discomfort | After each of the 12 training sessions, twice a week for 6 weeks
  Category Ratio Scale (0-10)
rating of thermal sensation | After each of the 12 therapy sessions, twice a week for 6 weeks
  9 point likert scale (4 / -4)
rating of perceived comfort | After each of the 12 therapy sessions, twice a week for 6 weeks
  5 point likert scale (0-4)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Clijsen, PhD, Principal Investigator — University of Applied Sciences and Arts of Southern Switzerland
Locations (1):
- University of Applied Sciences and Arts of Southern Switzerland, Landquart, Kanton Graubünden, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT06852872/Prot_SAP_001.pdf